CLINICAL TRIAL: NCT02944409
Title: Prospective Non-interventional, Prospective Multicenter Study of VEGA System® Prosthesis in the Total Knee Arthroplasty
Brief Title: VEGA System® Study in the Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1511
Record Dates: First submitted 2016-10-12; First posted 2016-10-25 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: total knee prothesis VEGA System — total knee replacement

SUMMARY:
This post-market clinical follow-up study intends to investigate long-term functionality of the VEGA System®. The design of the VEGA System® is meant to provide the patient with more knee mobility compared to their pre-operative state.The endpoint is the revision of at least one of the prosthesis components

ELIGIBILITY:
Inclusion Criteria

1. Patient from 18 to 75 years old
2. Patient is able to comply with follow-up requirements including postoperative self-evaluations.
3. Patient requires a primary knee replacement.
4. Patient has a diagnosis of osteoarthritis
5. Patient has intact collateral ligaments.

Exclusion Criteria

1. Vulnerable patient under legal protection
2. Patients with inflammatory arthritis.
3. Patients that have had a high tibial osteotomy or femoral osteotomy.
4. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Person for whom a replacement of knee was planed and for whom the surgeon planed to use VEGA System for the Knee Arthroplasty
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Survival rate of the prosthesis at 5 years | needs of revision of at least one of the prosthesis component evaluated 5 years after the knee arthroplasty
  If a patient withdraws from the study for any reason, counts as the end date for the survival of the implant of the last day on which the implants were well known even in place

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Privé des Bonnettes-Service de Chirurgie Orthopédique et Traumatologie, Arras
  - Hôpital Lariboisière- Service de Chirurgie Orthopédique et Traumatologie, Paris

IPD SHARING:
Plan to Share IPD: No